CLINICAL TRIAL: NCT04701853
Title: Specific Training After Stoma Surgery
Acronym: STASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FoU in VGR: 275326
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Colon Cancer
Keywords: Hernia; Abdominal muscles; Stabilizing training
MeSH Terms: conditions — Colonic Neoplasms; Hernia

STUDY DESIGN:
Intervention Model Description: A single blind, randomized, controlled, intervention study. Evaluation of the addition of specific muscle training for patients undergoing intestine surgery including a sigmoidostomy compared to standard care
Who Masked: Outcomes Assessor
Masking Description: Assessor will not be aware of which group the patients are included in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific abdominal muscle training (Experimental): Specific abdominal muscle training which is introduced preoperatively and performed the first year after surgery
  Interventions: Other: Specific abdominal muscle training
- Usual care treatment (Active Comparator): No specific abdominal muscle training
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Specific abdominal muscle training — Specific abdominal muscle training
  Arms: Specific abdominal muscle training
Other: Usual care — Care according to each center.
  Arms: Usual care treatment

SUMMARY:
In Sweden, approximately 43,000 people have undergone surgery with ileo-, colo- or urostomy. The most common type of stomy is a sigmoidostomy. A large proportion, about 50%, of patients who receive a permanent sigmoidostomy develop a parastomal hernia which may have major impact.

There are indications that specific abdominal exercise may reduce the risk of parastomal hernias, but randomized studies are lacking.

The aims of the study are:

1. to evaluate the effect of specific exercise to counteract the development of parastomal hernia in sigmoidostomy and the hernia's impact on ostomy function, physical function and quality of life.
2. to examine patients' experience of living with parastomal hernia. The study plans to include 240 patients who on will undergo surgery and receive a sigmoidostomy. These will be randomized to receive only advice according to the usual routine to avoid the development of parastomal hernia or these advice with the addition of specific abdominal muscle training. The training is initiated before the operation and is then carried out during the first postoperative year. Follow-up will be done with a clinical assessment and with measurement of bulge and size of the parastomal hernia manually, with electronic measuring equipment and via computed tomography images. Patients will assess their stoma and stoma function and assess any discomfort and its consequences of hernia via a study-specific questionnaire. Type of ostomy bandage will also be registered. The evaluation will be carried out 6, 12 and 36 months postoperatively.

Prior to the start of sub-study a, the planned measurement methods to assess whether a parastomal hernia is present will be tested for validity. In addition, a group of patients (≥15 people) with parastomal hernia will be included in a qualitative sub-study where they will be interviewed about their experiences of the hernia hernia and how it may affect daily life.

The present study will be able to answer whether specific exercise can reduce the risk of parastomal hernia. Methods for clinically assessing and evaluating bulging and hernias will be tested and evaluated in relation to patient-reported symptoms. In addition, the study will provide information about the patient's experience of having a parastomal hernia and how it affects daily life and physical activity. The results will provide an increased understanding of parastomal hernias, which may change the follow-up of patients in the future.

ELIGIBILITY:
Inclusion Criteria:

- A consecutive series of patients who are scheduled to have a permanent sigmoidostomy

Exclusion Criteria:

* Not Swedish speaking
* Impaired cognitive ability
* Physical disability that limits the possibility of carrying out the intervention.
* Lung disease including chronic cough.
* Previous hernia in the abdominal wall.
* Previous open abdominal surgery with scars ≥20 cm
* Spread malignant disease at inclusion
* Acute surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Parastomal hernia verified by computer tomography | 6 to 36 months after surgery
  Number of verified parastomal hernia by computer tomography

SECONDARY OUTCOMES:
Manual evaluation of parastomal hernia | 6 to 36 months after surgery
  Visual evaluation of parastomal hernia assessed by Yes/No/Unsure
Measurement of parastomal hernia | 6 to 36 months after surgery
  Size of the hernia by caliper and app
Stomal function- symptoms | 6 to 36 months after surgery
  Questionnaire including stomal function, by Smietanski. 15 items answered by Likert scales from 0 (no symptoms) to 10 (worst imaginable symptoms)
Stomal function in daily life | 6 to 36 months after surgery
  Questionnaire including stomal function in normal life, by Hjortswang 2006. Four questions which are answered by 6-levels Lickert scales from no (0) tom maximal (5) symptoms.
Generic Quality of life | 6 to 36 months after surgery
  EQ-5D Swedish version. 5 questions where lower scores indicate higher quality of life.
Stoma specific Quality of Life | 6 to 36 months after surgery
  Stoma-QoL by Kald et al 2009. 20 questions with answers from 1 (always) to not at all (4).
Physical activity level | Preoperatively to 36 months after surgery
  Grimby Scale, A scale from 1-6 where a higher score indicates higher level of physical activity
Back pain | Preoperatively to 36 months after surgery
  Back pain questionnaire by Granström et al 2020. Includes two visual analogue scales from 0 (no pain ) to 100 (Worst imaginable pain) mm and six questions which are answered on a Likert scale (4-5 levels) from no to maximal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Fagevik Olsén, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (4):
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Helsingborgs lasarett, Helsingborg
  - Örebro Universitetssjukhus, Örebro
  - Skövde Sjukhus, Skövde

IPD SHARING:
Plan to Share IPD: Undecided